CLINICAL TRIAL: NCT04950712
Title: A Descriptive, Prospective, Multi-country, Multicentre Study to Assess Performance of Genital Herpes Simplex Virus-2 (HSV-2) Related Disease Endpoints Based on Patient-reported Health Outcomes, Self-swabbing Collected Via Decentralised Approach in Patients ≥ 18 Years of Age in the United States and Europe.
Brief Title: An Epidemiological Study to Assess Performance of Using Healthcare Tools to Understand Genital Herpes Simplex Virus-2 (HSV-2) in Patients ≥ 18 Years of Age in the United States and Europe.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 214523
Record Dates: First submitted 2021-06-09; First posted 2021-07-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Herpes Genitalis
Keywords: Herpes Simplex Virus-2; HSV-2 genital herpes; HSV-2 recurrence
MeSH Terms: conditions — Herpes Genitalis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Overall Study Group: Patients aged 18 years old or above, with HSV-2 genital herpes, who are recruited in specific community settings in the United States and in Europe.
  Interventions: Procedure: Blood sampling; Procedure: Anogenital lesion swab collection

INTERVENTIONS:
Procedure: Blood sampling — Blood samples for HSV-2 testing and for HIV test are collected from patients at screening visit (first visit).
Procedure: Anogenital lesion swab collection — Anogenital lesion swab of all lesions are collected at screening visit (only for newly infected HSV-2 patients) and at first genital HSV-2 recurrence during the study period.

SUMMARY:
The aim of this study is to assess performance of using healthcare tools to understand genital Herpes Simplex Virus-2 (HSV-2) in patients ≥ 18 years of age in the United States and Europe.

More specifically, the study aims to evaluate patient-reported outcome and quality-of-life endpoints as well as the performance study procedures in a decentralised setting. Ultimately, this study will allow generating additional real-world evidence (RWE) on patterns of recurrences and other key parameters.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥18 years old.
* Written informed consent obtained from the patient prior to performance of any study-specific procedure.
* History of at least one episode of HSV-2 genital herpes lesions in the 12 months preceding the screening, and seropositive for HSV-2 as determined by Western blot OR PCR-positive for HSV-2 (newly diagnosed patients).
* Patients who are medically stable in the opinion of the investigator.
* Patients who, in the opinion of the investigator, are able to understand and comply with the study requirements (attend regular telephone calls/study site visits/home visits/self-completion of questionnaires, self-swabbing).
* Seronegative for HIV, as determined by laboratory testing. Patients documented to be positive to HIV will not be eligible for study participation

Exclusion Criteria:

* Prior receipt of a vaccine or candidate vaccine containing HSV antigens.
* Immunocompromised patients, as per medical history and investigator judgement.
* Other genital tract disorders or sexually transmitted diseases that may interfere with the assessment of the study (as per investigator's judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in specific community settings in the United States and in Europe. Screening logs will be used to assess participation rate.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with Polymerase Chain Reaction (PCR)-confirmed genital HSV-2 recurrences | During the 2-year follow-up period (from Enrolment Visit at Day 1 up to Month 24)
  Genital HSV-2 recurrence is defined as presence of lesions in anogenital area (swelling, blisters, sores, crusts) and, a positive HSV-2 PCR test.
Duration of PCR-confirmed genital HSV-2 recurrences | During the 2-year follow-up period (from Enrolment Visit at Day 1 up to Month 24)
  Duration of a recurrence is defined as number of consecutive days with the presence of HSV-2 lesion(s) and associated prodromal symptoms and/or erythema (skin redness).

SECONDARY OUTCOMES:
Change in severity of symptoms during HSV-2 genital herpes recurrence assessed by Patient global impression of severity (PGI-S) questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Change in severity of symptoms during HSV-2 genital herpes recurrence assessed by Patient global impression of change (PGI-C) questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Change in severity of symptoms during HSV-2 genital herpes recurrence assessed by Herpes symptoms checklist (HSC) questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Change in severity of symptoms during HSV-2 genital herpes recurrence assessed by Herpes outbreak impact (HOIQ) questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Impact of HSV-2 genital herpes recurrence on patients' daily functioning and quality-of-life as assessed by HSC questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Impact of HSV-2 genital herpes recurrence on patients' daily functioning and quality-of-life as assessed by HOIQ questionnaire | From the onset of recurrence until the end of the episode, assessed throughout the study period (for approximately 24 months)
Impact of HSV-2 genital herpes recurrence on patients' daily functioning and quality-of-life as assessed by EuroQoL-5 dimension (EQ-5D) health questionnaire | At Enrolment Visit (Day 1) and at Day 1 of each PCR-confirmed recurrence
Long-term impact on the quality-of-life of patients with symptomatic HSV-2 genital herpes as assessed by Recurrent genital herpes quality-of-life (RGHQoL) questionnaire | At Enrolment Visit (Day 1) and every 3 months until study completion at Month 24
Long-term impact on the quality-of-life of patients with symptomatic HSV-2 genital herpes as assessed by short form-12 questionnaire | At Enrolment Visit (Day 1) and every 3 months until study completion at Month 24
Number of self-swabs collected during genital HSV-2 recurrences throughout the study period | Throughout the study period (from Day 1 up to Month 24)
HSV-2 PCR self-swab results | At first genital HSV-2 recurrence, assessed throughout the study period (for approximately 24 months)
HSV-2 PCR investigator swab results | At first genital HSV-2 recurrence, assessed throughout the study period (for approximately 24 months)
Number of patients reporting genital HSV-2 recurrences by using eDiary | Throughout the study period (from Day 1 up to Month 24)
Number of patients reporting genital HSV-2 recurrence during the 3 monthly calls with the investigator | Throughout the study period (from Day 1 up to Month 24)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- United States (19):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lawrenceville, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Richmond, Virginia
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
- France (6):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Toulouse
- Italy (4):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Roma
- Spain (6):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Valencia
- United Kingdom (6):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Leeds Yorkshire
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: No